CLINICAL TRIAL: NCT04774861
Title: Correlation of Cardiac Computed Tomography Angiography Dimensions and Ethnicity in Trinidad: The CADET Study
Brief Title: Correlation of Cardiac Computed Tomography Angiography Dimensions and Ethnicity in Trinidad
Acronym: CADET
Status: Completed | Type: Observational
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Naveen Seecheran, Co-Investigator, The University of The West Indies
Other Study IDs: CREC-SA.0451/08/2020
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CCTA Group: This is an all-comers group, of all ages and ethnicities who have been evaluated with a CCTA from 2017-2020.

SUMMARY:
The aim of this study is to compare coronary artery dimensions on Cardiac CT angiography amongst different ethnicities in Trinidad.

DETAILED DESCRIPTION:
The aim of this study is to compare coronary artery dimensions on Cardiac CT angiography amongst different ethnicities in Trinidad.

ELIGIBILITY:
Inclusion Criteria:

1. CCTA for chest pain
2. All ethnicities
3. All genders

Exclusion Criteria:

1. Patients who did not provide consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient who underwent CCTA from 2017-2020 at the Eric Williams Medical Sciences Complex.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Coronary Artery Dimension | 2 years
  Coronary Artery Dimension of proximal, middle and distal LAD, LCx and RCA

CONTACTS AND LOCATIONS:
Locations (1):
- The University of the West Indies, Saint Augustine, North, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: Yes
All materials will be made available for sharing.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 5 years.
Access Criteria: A written request to Study Team.

REFERENCES:
- [Derived] Welch T, Rampersad F, Motilal S, Seecheran NA. Comparison of cardiac CT angiography coronary artery dimensions and ethnicity in Trinidad: the CADET pilot study. Open Heart. 2022 Mar;9(1):e001922. doi: 10.1136/openhrt-2021-001922. PMID 35354659